CLINICAL TRIAL: NCT03792750
Title: A Phase 1/2 Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of BMS-986205 Alone and in Combination With Nivolumab in Chinese Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of BMS-986205 Alone and in Combination With Nivolumab in Chinese Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA017-076
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — linrodostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Arm A (Experimental): 2 week BMS-986205 monotherapy lead in followed by BMS-986205 + Nivo combination therapy
  Interventions: Drug: BMS-986205; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986205 — Specified Dose on Specified Day
Biological: Nivolumab — Specified Dose on Specified Day
  Other Names: BMS-936558

SUMMARY:
The purpose of this study is to determine safety and effectiveness of experimental medication BMS-986205 in combination with Nivolumab in patients with cancers that are advanced or have spread.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic or cytological confirmation of a solid tumor that is advanced with measureable disease per RECIST v1.1
* Participants must have received, and then progressed or been intolerant to at least one standard treatment regimen in the advanced or metastatic setting
* Participants must have an ECOG performance status of less than or equal to 1
* Participants must have at least 1 lesion with measurable disease as defined by RECIST Version 1.1

Exclusion Criteria:

* Participants must not have suspected, known, or progressive CNS metastases, have untreated CNS metastases, or have the CNS as the only site of disease
* Participants with prior exposure to anti PD-1 or anti-PDL1 therapy
* Participants must not have a history of allergy to any of the study treatment components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-31 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Individual patient level data from this study may be shared with qualified researchers, upon request, following the timelines and process detailed on https://www.bms.com/researchers-and-partners/independent-research/data-sharing-request-process.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-986205 in Combination With Nivolumab: Study treatment starts with a monotherapy therapy 2-week lead-in treatment (Cycle 0) consisting of a single oral daily dose of 100 mg BMS-986205. Followed by combination therapy cycles comprised of an oral daily dose of 100mg BMS-986205 and one dose of 480mg nivolumab administered intravenously Q4W on Day 1 of each treatment cycle up to 12 cycles.
Period: Overall Study
Arm/Group | BMS-986205 in Combination With Nivolumab
Started | 12
Completed | 9
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 12

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Adverse Events (AE)
Description: The number of participants experiencing adverse events (AEs) to assess the safety and tolerability of BMS-986205.
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 2 years)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants | 11

2. Primary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAE)
Description: The number of participants experiencing serious adverse events (SAEs) to assess the safety and tolerability of BMS-986205
  Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 2 years)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants | 3

3. Primary Outcome: The Number of Participants Experience Adverse Events (AE) Leading to Discontinuation
Description: The number of participants experiencing adverse events (AEs) leading to discontinuation to assess the safety and tolerability of BMS-986205
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 2 years)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants | 5

4. Primary Outcome: Number of Participant Deaths
Description: The number of participants who died in each arm during the study to assess the safety and tolerability of BMS-986205.
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 2 years)
Population: All treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants | 3

5. Primary Outcome: The Number of Participants Experiencing Laboratory Abnormalities in Specific Liver Tests
Description: The number of participants with clinical laboratory test abnormalities in specific liver tests based on US conventional units to assess the safety and tolerability of BMS-986205.
  The number of participants with the following laboratory abnormalities will be summarized:
  ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN Total bilirubin > 1.5 x ULN and 2 x ULN Concurrent (within 1 day) ALT or AST > 3 x ULN with total bilirubin > 2 x ULN Concurrent (within 30 days) ALT or AST > 3 x ULN with total bilirubin > 2 x ULN
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 2 years)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants
  ALT OR AST > 3XULN | 3
  ALT OR AST> 5XULN | 2
  ALT OR AST> 10XULN | 0
  ALT OR AST > 20XULN | 0
  TOTAL BILIRUBIN > 1.5XULN | 2
  TOTAL BILIRUBIN > 2XULN | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0

6. Primary Outcome: The Number of Participants Experiencing Laboratory Abnormalities in Specific Thyroid Tests
Description: The number of participants with clinical laboratory test abnormalities based on US conventional units to assess the safety and tolerability of BMS-986205.
  The number of subjects with the following laboratory abnormalities will be summarized:
  TSH > ULN WITH TSH <= ULN AT BASELINE WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN (Within a 2-week window after the abnormal TSH test date) WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN (Within a 2-week window after the abnormal TSH test date) WITH FT3/FT4 TEST MISSING (Within a 2-week window after the abnormal TSH test date) TSH < LLN WITH TSH >= LLN AT BASELINE WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN (Within a 2-week window after the abnormal TSH test date) WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN (Within a 2-week window after the abnormal TSH test date) WITH FT3/FT4 TEST MISSING (Within a 2-week window after the abnormal TSH test date)
Time Frame: From first dose to 100 days after last dose of study therapy (up to approximately 2 years)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants
  TSH > ULN | 4
  TSH > ULN WITH TSH <= ULN AT BASELINE | 4
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 2
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 4
  TSH > ULN WITH FT3/FT4 TEST MISSING | 0
  TSH < LLN | 5
  TSH <LLN WITH TSH >= LLN AT BASELINE | 4
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 0
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 5
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0

7. Primary Outcome: (Cmax) Maximum Observed Plasma Concentration
Description: The maximum observes plasma concentration was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 days 1, 14, Cycle 1 day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
ng/mL
  C0D1 | 596.0 (44.138)
  C0D14 | 701.9 (24.870)
  C1D1 | 781.0 (18.933)

8. Primary Outcome: (Tmax) Time of Maximum Observed Plasma Concentration
Description: The time of maximum observed plasma concentration was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 days 1, 14, Cycle 1 day 1
Population: Evaluable PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
hours
  C0D1 | 2.5 [1 to 3]
  C0D14 | 2.5 [2 to 4]
  C1D1 | 2.5 [1.1 to 4]

9. Primary Outcome: (AUC(TAU)) Area Under the Concentration-time Curve in One Dosing Interval
Description: The area under the concentration-time curve in one dosing interval was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 days 1, 14, Cycle 1 day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
ng*h/mL
  C0D1 | 3380.8 (34.754)
  C0D14 | 6048.3 (38.830)
  C1D1 | 5922.3 (32.572)

10. Primary Outcome: (CLT/F) Apparent Total Body Clearance
Description: The apparent total body clearance was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 day 14, Cycle 1 day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
L/h
  CYCLE0 DAY14 | 16.5 (38.830)
  CYCLE1 DAY1 | 16.9 (32.572)

11. Primary Outcome: (T-HALF (Eff, AUC)) Effective Elimination Half-life
Description: The effective elimination half-life was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab. T-HALF (eff, AUC) explains the degree of AUC accumulation observed.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 day 14
Population: Evaluable PK Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 11
Hours | 22.9 (9.40)

12. Primary Outcome: (AI_CMAX) Accumulation Index
Description: The accumulation index was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab. AI is calculated based on ratio of Cmax at steady state to after the first dose.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 day 14
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
ng/mL | 1.2 (42.479)

13. Primary Outcome: (AI_AUC ) Accumulation Index
Description: The accumulation index was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab. AI is calculated based on ratio of AUC(TAU) at steady state to after the first dose.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 day 14
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
ng*h/mL | 1.8 (32.866)

14. Primary Outcome: (Ctrough) Trough Observed Plasma Concentration
Description: The trough observed plasma concentration was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 day 2, 8, 14, Cycle 1 day 1, 2, Cycle 3, 5, 9, 13, and 17 day 1
Population: Evaluable PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 12
ug/mL
  Cycle0 Day2 | 51.2 (35.255)
  Cycle0 Day8 | 117.4 (44.282)
  Cycle0 Day14 | 154.9 (51.005)
  Cycle1 Day1 | 141.5 (60.276)
  Cycle1 Day2 | 150.2 (46.971)
  CYCLE3 DAY1: number analyzed (Participants) | 5
  CYCLE3 DAY1 | 161.3 (97.305)
  CYCLE5 DAY1: number analyzed (Participants) | 4
  CYCLE5 DAY1 | 239.2 (38.883)
  CYCLE9 DAY1: number analyzed (Participants) | 2
  CYCLE9 DAY1 | 144.0 (64.086)
  CYCLE13 DAY1: number analyzed (Participants) | 1
  CYCLE13 DAY1 | 134.0 (NA) — Coefficient of Variation is not evaluable for only 1 participant
  CYCLE17 DAY1: number analyzed (Participants) | 1
  CYCLE17 DAY1 | 3.2 (NA) — Coefficient of Variation is not evaluable for only 1 participant

15. Primary Outcome: (percentUR24) Percent Urinary Recovery Over 24 Hours
Description: The percent urinary recovery over 24 hours was collected to characterize the pharmacokinetics of BMS-986205 administered alone and in combination with nivolumab.
  BMS-986205 had minimal evaluable concentration in urine to derive the parameter.
Time Frame: pre-dose, 1, 2, 3, 4, 6, 8 hours post dose on Cycle 0 Day 1 and 2
Population: Evaluable PK Population
Arm/Group | BMS-986205 in Combination With Nivolumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the total number of participants whose best overall response (BOR) is either a completer response (CR) or partial response (PR) divided by the total number of participants in the population of interest. Assessed per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 by investigator
  BOR is defined as the best response designation over the study as a whole, recorded between the dates of first dose until the last tumor assessment prior to subsequent therapy.
Time Frame: From first dose up to approximately 2 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Groups:
- BMS-986205 Monotherapy and in Combination With Nivolumab: The treatment phase consists of the 2-week monotherapy lead-in (Cycle 0) and up to twelve 4-week combination therapy cycles. The 2-week lead-in treatment consists of a single oral daily dose of BMS-986205. The combination therapy cycles are comprised of an oral daily dose of BMS-986205 and one dose of nivolumab administered intravenously Q4W on Day 1 of each treatment cycle up to 12 cycles. Total study treatment period is up to 50 weeks
Arm/Group | BMS-986205 Monotherapy and in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants | 1

17. Secondary Outcome: Best Overall Response (BOR)
Description: BOR defined as the best response designation over the study as a whole, recorded between the dates of first dose until the last tumor assessment prior to subsequent therapy. Assessed per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 by investigator
Time Frame: From first dose up to approximately 2 years
Population: All treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 Monotherapy and in Combination With Nivolumab
Number analyzed (Participants) | 12
Participants
  COMPLETE RESPONSE (CR) | 0
  PARTIAL RESPONSE (PR) | 1
  STABLE DISEASE (SD) | 5
  PROGRESSIVE DISEASE (PD) | 5
  UNABLE TO DETERMINE (UTD) | 1

18. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) is defined as the time between the date of first response and the date of disease progression or death, whichever occurs first. Assessed per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 by investigator.
Time Frame: From first dose up to approximately 2 years
Population: All treated participants with a BOR of CR or PR
Measure: Number; unit: Weeks
Arm/Group | BMS-986205 Monotherapy and in Combination With Nivolumab
Number analyzed (Participants) | 1
Weeks | 72

19. Secondary Outcome: Measurement of Serum Kynurenine Levels
Description: Measurement of kynurenine levels were assessed to characterize the pharmacodynamic activity of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: Baseline, pre-dose (C1D1), 6 hours post dose (C1D1), pre-dose (C1D2), and at disease progression (actually collected on C3D1, C6D1, C8D1, and end of treatment-an average of 12 cycles)
Population: All Treated Participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BMS-986205 Monotherapy and in Combination With Nivolumab
Number analyzed (Participants) | 12
ng/mL
  BASELINE | 189.6 (64.46)
  CYCLE 1 D1 6 HOUR POST-DOSE | 150.8 (45.39)
  CYCLE 1 D2 | 180.6 (49.33)
  CYCLE 3 D1: number analyzed (Participants) | 1
  CYCLE 3 D1 | 273.0 (NA) — SD is not applicable for 1 evaluable participant
  CYCLE 6 D1: number analyzed (Participants) | 1
  CYCLE 6 D1 | 111.0 (NA) — SD is not applicable for 1 evaluable participant
  CYCLE 8 D1: number analyzed (Participants) | 1
  CYCLE 8 D1 | 124.0 (NA) — SD is not applicable for 1 evaluable participant
  END OF TREATMENT: number analyzed (Participants) | 2
  END OF TREATMENT | 198.5 (50.2)

20. Secondary Outcome: Measurement of Tryptophan Levels
Description: Measurement of tryptophan levels were assessed to characterize the pharmacodynamic activity of BMS-986205 administered alone and in combination with nivolumab.
Time Frame: as for outcome 19
Population: All Treated Participants
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BMS-986205 Monotherapy and in Combination With Nivolumab
Number analyzed (Participants) | 12
ng/mL
  BASELINE | 13445.8 (2671.18)
  CYCLE 1 D1 6 HOUR POST-DOSE | 14528.3 (2461.75)
  CYCLE 1 D2 | 12508.3 (2461.30)
  CYCLE 3 D1: number analyzed (Participants) | 1
  CYCLE 3 D1 | 17900.0 (NA) — SD is not applicable for 1 evaluable participant
  CYCLE 6 D1: number analyzed (Participants) | 1
  CYCLE 6 D1 | 13200.0 (NA) — SD is not applicable for 1 evaluable participant
  CYCLE 8 D1: number analyzed (Participants) | 1
  CYCLE 8 D1 | 13200.0 (NA) — SD is not applicable for 1 evaluable participant
  END OF TREATMENT: number analyzed (Participants) | 2
  END OF TREATMENT | 14200.0 (3394.11)

21. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to Nivolumab
Description: The number of participants with positive or negative anti-drug antibodies (ADA) to nivolumab was collected to characterize the immunogenicity of nivolumab when administered in combination with BMS-986205.
  Baseline ADA Positive: A subject with baseline ADA-positive sample. ADA Positive: A subject with at least one ADA-positive sample relative to baseline.
  Neutralizing Positive: At least one ADA-positive sample with neutralizing antibodies detected post-baseline ADA Negative: A subject with no ADA-positive sample after initiation of treatment.
Time Frame: Baseline, pre-dose (C1D1, C3D1, every 4 Cycles from C5D1), end of treatment - an average of 12 cycles, and follow up. (up to approximately 2 years)
Population: All Nivolumab Treated Subjects with Baseline and at Least One Post-Baseline Immunogenicity Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986205 Monotherapy and in Combination With Nivolumab
Number analyzed (Participants) | 7
Participants
  BASELINE ADA POSITIVE | 1
  ADA POSITIVE | 0
  NEUTRALIZING POSITIVE | 1
  ADA NEGATIVE | 7

ADVERSE EVENTS:
Time Frame: First dose and 100 days after last dose of study therapy (Up to approximately 2 years)
Arm/Group | BMS-986205 in Combination With Nivolumab
All-Cause Mortality (participants affected / at risk) | 3/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986205 in Combination With Nivolumab (N=12)
Tuberculosis (Infections and infestations) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986205 in Combination With Nivolumab (N=12)
Anaemia (Blood and lymphatic system disorders) | 9
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Uveitis (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 8
Blood alkaline phosphatase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 4
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
C-reactive protein increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Myoglobin blood increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Thyroxine increased (Investigations) | 1
Weight decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Dizziness (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Leukoderma (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT03792750/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT03792750/SAP_001.pdf